CLINICAL TRIAL: NCT01704378
Title: A Multi-National, Multi-Centre, Open-Labelled Extension Study Assessing the Long-Term Safety of Biphasic Insulin Aspart 30 in NovoMix®30 FlexPen™ in Type 2 Diabetic Patients Previously Treated in BIAsp-1236
Brief Title: Efficacy and Safety of Biphasic Insulin Aspart 30 FlexPen™ in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1386
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIAsp (Experimental)
  Interventions: Drug: biphasic insulin aspart

INTERVENTIONS:
Drug: biphasic insulin aspart — Individually adjusted dose. Injected subcutaneously (s.c., under the skin) twice daily before breakfast and evening meal

SUMMARY:
This trial is conducted in Europe. The aim of this trial investigate the the long-term safety of biphasic insulin aspart 30 in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any trial-related activities
* Completed the trial BIAsp-1236

Exclusion Criteria:

* Planned changes in use of any prescription medication that may interfere with glucose regulation
* Known or suspected allergy to trial products or related products
* Women who are having the intention of becoming pregnant, or are judged not to be using adequate contraceptive measures
* Any other significant condition or concomitant disease or any condition that would interfere with participation as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2001-04-18 (Actual); Primary Completion 2003-03-14 (Actual); Study Completion 2003-03-14 (Actual)

PRIMARY OUTCOMES:
Number of Hypoglycaemic episodes
Occurrence of adverse events

SECONDARY OUTCOMES:
HbA1c (glycosylated haemoglobin)
Prandial increment in blood glucose
7-point blood glucose profile

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (17):
- Finland (3):
  - Novo Nordisk Investigational Site, Kotka
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Lahti
- Norway (5):
  - Novo Nordisk Investigational Site, Gjøvik
  - Novo Nordisk Investigational Site, Horten
  - Novo Nordisk Investigational Site, Kirkenær
  - Novo Nordisk Investigational Site, Kongsvinger
  - Novo Nordisk Investigational Site, Notodden
- Sweden (3):
  - Novo Nordisk Investigational Site, Falun
  - Novo Nordisk Investigational Site, Helsingborg
  - Novo Nordisk Investigational Site, Motala
- United Kingdom (6):
  - Novo Nordisk Investigational Site, Derby
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, Scarborough
  - Novo Nordisk Investigational Site, Wirral, Merseyside

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com